CLINICAL TRIAL: NCT03581279
Title: Detection of Borrelia Bacteria in Early Stage Lyme Borreliosis Using the T2Lyme Panel
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment levels insufficient to continue.
Sponsor: T2 Biosystems (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: PRO-000879
Record Dates: First submitted 2018-06-26; First posted 2018-07-10 (Actual); Results first posted 2022-01-31 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Lyme Disease
MeSH Terms: conditions — Lyme Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All patients are assigned a unique study ID number to de-identify them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- EM present (Active Comparator): All patients must display signs/symptoms of Lyme disease as well as exhibit an EM lesion.
  Interventions: Device: T2Lyme Panel testing
- No EM present (Active Comparator): All patients must display signs/symptoms of Lyme disease but do not have an EM lesion.
  Interventions: Device: T2Lyme Panel testing

INTERVENTIONS:
Device: T2Lyme Panel testing — The T2Lyme Panel is an investigational use in vitro diagnostic (IVD) designed to qualitatively detect and identify the major causative agents of Lyme disease (Borrelia burgdorferi, Borrelia afzelii, Borrelia garinii, as well as an inclusive Borrelia spp. detection channel) from K2EDTA human whole blood samples.

SUMMARY:
The T2Lyme assay will be compared to Borrelia culture from erythema migrans (EM) biopsy and/or detection of the C6 antigen in serum collected prospectively from patients suspected of early Lyme disease.

DETAILED DESCRIPTION:
The objective of this study is to demonstrate the clinical performance of the T2Lyme Panel on the T2Dx instrument. The assay will be compared to Borrelia culture from erythema migrans (EM) biopsy and/or detection of the C6 antigen in serum collected prospectively from patients suspected of early Lyme disease. The data from this study will be used to support a de novo application for the T2Lyme Panel to the U.S. Food and Drug Administration (FDA) for product approval.

The T2Lyme Panel is an investigational use in vitro diagnostic (IVD) designed to qualitatively detect and identify the major causative agents of Lyme disease (Borrelia burgdorferi, Borrelia afzelii, Borrelia garinii, as well as an inclusive Borrelia spp. detection channel) from K2EDTA human whole blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Presence of erythematous skin lesion, consistent with erythema migrans (EM).
* Age 18 or older.
* Ability to read, comprehend, and sign the informed consent form.
* Two (2) or more signs/symptoms of Lyme Disease

Exclusion Criteria:

* Subject has medically diagnosed bleeding disorder.
* Having had taken antibiotics in the past 30 days.
* EM located on face or neck.
* Unable to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - South County Internal Medicine, Wakefield, Rhode Island
  - Gundersen Health System, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No
No data will be shared

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EM Present | No EM Present
Started | 18 | 0
Completed | 16 | 0
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: The "No EM present" arm of this study was never initiated.
Groups:
- Total: Total of all reporting groups
Arm/Group | EM Present | No EM Present | Total
Number analyzed (Participants) | 18 | 0 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 0 | 8
  >=65 years | 10 | 0 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (12) |  | 66 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 14 | 0 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 0 |  | 0
  More than one race | 0 |  | 0
  Unknown or Not Reported | 18 |  | 18
Region of Enrollment [Number; unit: participants]
  United States | 18 |  | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Lyme Disease Detected in Human Whole Blood Samples
Description: Qualitative detection of genetic material (DNA) from the major causative agents of Lyme disease (Borrelia burgdorferi, Borrelia afzelii, Borrelia garinii, as well as inclusive Borrelia spp.) from K2EDTA human whole blood samples using the T2Dx instrument and T2Lyme reagents.
Time Frame: 1 day
Population: The "No EM present" arm of the study was never initiated.
Measure: Count of Participants; unit: Participants
Arm/Group | EM Present | No EM Present
Number analyzed (Participants) | 18 | 0
Participants | 18 | 0

ADVERSE EVENTS:
Time Frame: 45 - 60 days
Description: No participants were enrolled in the "no EM present" arm of the study.
Arm/Group | EM Present | No EM Present
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/0
Other Adverse Events (participants affected / at risk) | 0/18 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT03581279/Prot_001.pdf